CLINICAL TRIAL: NCT00004981
Title: A Phase IIIB Randomized, Multicenter Study of the Efficacy and Safety of Combivir 1 Tablet Po Bid Plus Ziagen 300mg Po Bid Versus an Abacavir 300mg/Lamivudine 150mg/Zidovudine 300mg Combination Tablet Po Bid, Administered for 24 Weeks in Subjects With HIV-1 Infection
Brief Title: Safety and Effectiveness of Three Anti-HIV Drugs Combined in One Pill (Trizivir)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 308A; ESS40005
Record Dates: First submitted 2000-03-13; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-06

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; Drug Administration Schedule; Lamivudine; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Combivir; abacavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Lamivudine; Zidovudine; lamivudine, zidovudine drug combination

INTERVENTIONS:
Drug: Abacavir sulfate, Lamivudine and Zidovudine
Drug: Lamivudine/Zidovudine
Drug: Abacavir sulfate

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of a pill called Trizivir that is a combination of three anti-HIV drugs (zidovudine, lamivudine, and abacavir). Zidovudine and lamivudine are often given combined in one pill (Combivir). In this study, Trizivir will be compared to Combivir plus abacavir.

DETAILED DESCRIPTION:
Patients are randomized to receive either the triple combination tablet (Trizivir) or to receive Combivir plus abacavir as a separate tablet. Patients take their study medications for 24 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 18 years old.
* Are HIV-positive.
* Are currently receiving one of the following anti-HIV drug combinations: Combivir plus abacavir, Combivir plus abacavir plus a protease inhibitor, or Combivir plus abacavir plus a non-nucleoside reverse transcriptase inhibitor (NNRTI). Patients must have been taking this drug combination for at least the past 16 weeks. This also must be the first anti-HIV drug combination the patient has received.
* Have a viral load (level of HIV in the blood) less than or equal to 400 copies/ml.
* Have CD4+ cell count greater than 200 cells/mm3.
* Agree to use effective methods of birth control.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have been diagnosed with AIDS.
* Have a gastrointestinal disorder that makes it difficult for patients to absorb food or to take medications by mouth.
* Have hepatitis.
* Have a serious medical condition, such as diabetes, congestive heart failure, or other heart disease.
* Are allergic to any of the study drugs.
* Abuse alcohol or drugs.
* Will not be available for the entire 24-week study period.
* Are pregnant or breast-feeding.
* Have taken or will need to take certain medications, including radiation therapy, chemotherapy, drugs that affect the immune system (such as interleukin), an HIV vaccine, foscarnet, and hydroxyurea.
* Are enrolled in another experimental drug study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - AIDS Healthcare Foundation, Los Angeles, California
  - Tower Infectious Disease Med Ctr, Los Angeles, California
  - Robert Scott MD, Oakland, California
  - St Lukes Medical Group, San Diego, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Specialty Med Care Ctrs of South Florida Inc, Miami, Florida
  - Saint Josephs Comprehensive Research Institute, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - New England Med Ctr, Boston, Massachusetts
  - Research Med Ctr, Kansas City, Missouri
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - St Luke Roosevelt Hosp, New York, New York
  - Lehigh Valley Hosp, Allentown, Pennsylvania
  - Hahnemann Univ Hosp, Philadelphia, Pennsylvania
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Burnside Clinic, Columbia, South Carolina
  - Univ of Tennessee, Memphis, Tennessee
  - Nashville Health Management Foundation / Vanderbilt Univ, Nashville, Tennessee
  - Nicholas Bellos, Dallas, Texas
  - Univ of Texas Med Branch, Galveston, Texas
  - Therapeutic Concepts, Houston, Texas